CLINICAL TRIAL: NCT05279430
Title: Effects of Inspiratory Muscle Training on Maximal Functional Capacity in Patients With Chronic COVID After Hospital Discharge
Brief Title: Effects of IMT on Functional Capacity in Patients With Chronic COVID After Hospital Discharge
Acronym: InsCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Patricia Palau, Principal Investigator and clinical professor, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/226
Record Dates: First submitted 2022-03-12; First posted 2022-03-15 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients allocated to the control arm will not receive inspiratory muscle training. They will be checked each week by a physiotherapist responsible for training intervention who will measure their maximal inspiratory pressure
- Inspiratory muscle training (Active Comparator): Patients allocated to the IMT arm will be instructed to train at home twice daily, for 20 minutes each session, using a Threshold inspiratory muscle trainer (Respironics Inc., Parsippany, NJ). They will be instructed by a physiotherapist responsible for training intervention and educated to maintain diaphragmatic breathing during the training period. The subjects will start breathing at a resistance equal to 25% to 30% of their maximal inspiratory mouth pressure (MIP) for 1 week. The respiratory therapist will examine the patients at weekly intervals by checking the diary card and measuring the MIP each time. The resistance will be modified each session according to the 25% to 30% of their MIP measured.
  Interventions: Behavioral: Inspiratory muscle training

INTERVENTIONS:
Behavioral: Inspiratory muscle training — Patients allocated to the IMT arm will be instructed to train at home twice daily, for 20 minutes each session, using a Threshold inspiratory muscle trainer (Respironics Inc., Parsippany, NJ). They will be instructed by a physiotherapist responsible for training intervention and educated to maintain diaphragmatic breathing during the training period. The subjects will start breathing at a resistance equal to 25% to 30% of their maximal inspiratory mouth pressure (MIP) for 1 week. The respiratory therapist will examine the patients at weekly intervals by checking the diary card and measuring the MIP each time. The resistance will be modified each session according to the 25% to 30% of their MIP measured.
  Arms: Inspiratory muscle training

SUMMARY:
Exercise intolerance and fatigue are the most common symptoms in patients with chronic COVID after hospital discharge. Muscle deconditioning, dysautonomia, and exercise hyperventilation have been proposed as potential mechanisms contributing to exercise functional capacity limitation in Long-COVID. Along this line, combined exercise training or inspiratory muscle training (IMT) alone have already been demonstrated to be feasible therapeutic options for Long-COVID patients. However, we do not have evidence about the effects of a home-based IMT program for 12-week on peak oxygen consumption (peakVO2). in patients chronic COVID (>3 months) after hospital discharge.

This is a prospective study, blinded for the evaluator, randomized (1:1) to receive standard management alone or combined with a program of IMT that will be carried out in a single center. After randomization, patients will be clinically evaluated. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing (CPET) at 12-week. Patients with chronic COVID (>3 months) after hospital discharge will be enrolled. A sample size estimation [alfa: 0.05, power: 80%, a 15% loss rate, and at least a delta change of mean peakVO2: +3 mL/kg/min (SD±2.5)] of 26 patients (13 per arm) would be necessary to test our hypothesis.

DETAILED DESCRIPTION:
Exercise intolerance and fatigue are the most common symptoms in patients with chronic COVID after hospital discharge. Muscle deconditioning, dysautonomia, and exercise hyperventilation have been proposed as potential mechanisms contributing to exercise functional capacity limitation in Long-COVID. Along this line, combined exercise training or inspiratory muscle training (IMT) alone have already been demonstrated to be feasible therapeutic options for Long-COVID patients. However, we do not have evidence about the effects of a home-based IMT program for 12-week on peak oxygen consumption (peakVO2). in patients chronic COVID (>3 months) after hospital discharge.

This is a prospective study, blinded for the evaluator, randomized (1:1) to receive standard management alone or combined with a program of IMT that will be carried out in a single center. Patients allocated to the IMT arm will be instructed to train at home twice daily, for 20 minutes each session, using a Threshold inspiratory muscle trainer (Respironics Inc., Parsippany, NJ). They will be instructed by a physiotherapist responsible for training intervention and educated to maintain diaphragmatic breathing during the training period. The subjects will start breathing at a resistance equal to 25% to 30% of their maximal inspiratory mouth pressure (MIP) for 1 week. The respiratory therapist will examine the patients at weekly intervals by checking the diary card and measuring the MIP each time. The resistance will be modified each session according to the 25% to 30% of their MIP measured. After randomization, patients will be clinically evaluated. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing (CPET) at 12-week. Patients with chronic COVID (>3 months) after hospital discharge will be enrolled. A sample size estimation [alfa: 0.05, power: 80%, a 15% loss rate, and at least a delta change of mean peakVO2: +3 mL/kg/min (SD±2.5)] of 26 patients (13 per arm) would be necessary to test our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic adult patients >18 years old with the previous admission due to SARS-CoV-2 pneumonia
2. > 3-month after discharge
3. The patient provides informed consent

Exclusion Criteria:

1. Inability to perform a maximal baseline exercise test
2. Structural heart disease, valve heart disease, or diastolic dysfunction estimated by 2-dimensional echocardiography
3. Patients with previous ischemic heart disease, heart failure, myocardiopathy, or myocarditis
4. Effort angina or signs of ischemia during CPET
5. Significant primary pulmonary disease, including a history of pulmonary arterial hypertension, chronic thromboembolic pulmonary disease, or chronic obstructive pulmonary disease

(g) Treatment with digitalis, calcium channel blockers, β-blocker or ivabradine (h) Patients with chronic kidney disease (glomerular filtration rate <60mL/min/1.73m2) (i) Patients with pacemakers or previous history of atrial fibrillation; (j) patients with autoimmune, inflammatory or active neoplastic disease k) Anemia (l) Pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption | 12-week
  Maximal functional capacity will be evaluated with incremental and symptom-limited cardiopulmonary exercise testing. Peak oxygen consumption (peakVO2) will be considered the highest value of VO2 during the last 20 seconds of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Palau, MD, PhD, Principal Investigator — INCLIVA-Hospital Clínico Universitario
Locations (1):
- INCLIVA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 3 months after publication
Access Criteria: Data is available upon the reasonable request

REFERENCES:
- [Result] Palau P, Dominguez E, Lopez L, Heredia R, Gonzalez J, Ramon JM, Serra P, Santas E, Bodi V, Sanchis J, Chorro FJ, Nunez J. Inspiratory Muscle Training and Functional Electrical Stimulation for Treatment of Heart Failure With Preserved Ejection Fraction: Rationale and Study Design of a Prospective Randomized Controlled Trial. Clin Cardiol. 2016 Aug;39(8):433-9. doi: 10.1002/clc.22555. Epub 2016 Aug 2. PMID 27481035
- [Result] Palau P, Dominguez E, Nunez E, Schmid JP, Vergara P, Ramon JM, Mascarell B, Sanchis J, Chorro FJ, Nunez J. Effects of inspiratory muscle training in patients with heart failure with preserved ejection fraction. Eur J Prev Cardiol. 2014 Dec;21(12):1465-73. doi: 10.1177/2047487313498832. Epub 2013 Jul 17. PMID 23864363
- [Derived] Palau P, Dominguez E, Gonzalez C, Bondia E, Albiach C, Sastre C, Martinez ML, Nunez J, Lopez L. Effect of a home-based inspiratory muscle training programme on functional capacity in postdischarged patients with long COVID: the InsCOVID trial. BMJ Open Respir Res. 2022 Dec;9(1):e001439. doi: 10.1136/bmjresp-2022-001439. PMID 36549786
- [Derived] Palau P, Dominguez E, Sastre C, Martinez ML, Gonzalez C, Bondia E, Albiach C, Nunez J, Lopez L. Effect of a home-based inspiratory muscular training programme on functional capacity in patients with chronic COVID-19 after a hospital discharge: protocol for a randomised control trial (InsCOVID trial). BMJ Open Respir Res. 2022 Jul;9(1):e001255. doi: 10.1136/bmjresp-2022-001255. PMID 35790316